CLINICAL TRIAL: NCT00373646
Title: Phase II Trial of Thalidomide (Thalidomide Pharmion) in Patients With Advanced or Relapsed Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT)
Brief Title: Thalidomide in Mucosa Associated Lymphoid Tissue (MALT) Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Medical University of Vienna, Dept of Internal Medicine I
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thalidomide-MALT; Eudract number 2005-000008-14
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: MALT Lymphoma
Keywords: MALT Lymphoma; thalidomide; disseminated MALT Lymphoma or at relapse following HP-eradication; or chemotherapy or radiation
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide, Pharmion — 200 mg p.o. daily

SUMMARY:
The purpose of this study is to evaluate Thalidomide for treatment of disseminated MALT Lymphoma or at relapse following helicobacter pylori (HP) - eradication or chemotherapy or radiation.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the effectivity and the safety of thalidomide in patients with disseminated MALT lymphoma or at relapse following HP-eradication, or chemotherapy or radiation. It is a phase II prospective single arm study with a target sample size of 16 patients. Thalidomide is given orally at an initial dose of 100 mg for a maximum duration of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed MALT lymphoma with measurable disease (Stage I-IV)
* With first or greater relapse after HP-eradication, radiation or chemotherapy
* Age > 18
* Must be able to tolerate therapy and have adequate cardiac, renal and hepatic function
* ECOG status _< 2
* Must be capable of understanding the purpose of the study and have given written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical potential of thalidomide to induce objective/histologic responses in patients with MALT lymphoma | 6 months

SECONDARY OUTCOMES:
To evaluate the safety of thalidomide in this patient population and to evaluate | 6 months
The impact of thalidomide on progression free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Raderer, Prof, Principal Investigator — Department of Internal Medicine I
Locations (1):
- Department of Internal Medicine I, Vienna, Austria